CLINICAL TRIAL: NCT05556772
Title: Estudio Oportunidad: Optimizing Screening for Cervical Cancer Among Women Living With HIV in the Dominican Republic
Brief Title: Optimizing Screening for Cervical Cancer Among Women Living With HIV in the Dominican Republic
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); US-Latin American-Caribbean HIV/HPV-Cancer Prevention Clinical Trials Network (ULACNet) (Unknown); Instituto Dermatológico Dominicano y Cirugía de Piel (IDCP) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: RG1122164; NCI-2021-14229 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1122164 (Other: Fred Hutch/University of Washington Cancer Consortium); ULACNET-302 (Other: DCP); U54CA242977 (NIH); 10893 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2022-08-29; First posted 2022-09-27 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Malignant Female Reproductive System Neoplasm
MeSH Terms: interventions — Specimen Handling; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (biospecimen collection, cytology, interview) (Experimental): Participants participate in an interview and clinical exam, lasting approximately 2 hours. Participants undergo vaginal self-sampling, cervical provider-sampling, and collection of blood and urine samples. Participants also undergo a pelvic exam. After first interview and clinical exam at enrollment, participants have two subsequent study visits over a 2 year period.
  Interventions: Procedure: Biospecimen Collection; Other: Interview

INTERVENTIONS:
Procedure: Biospecimen Collection — Collection of blood; urine; cervical, anal, vaginal samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection; Biopsy when indicated; Biological Sample Collected
Other: Interview — Attend interview

SUMMARY:
This study compares different screening approaches to detect abnormal cell growth on the cervix that could be an early sign of cervical cancer. The lesions are caused by an infection of human papillomavirus, also called HPV. Using new methods to detect HPV may help doctors find ways to improve cervical cancer screening for women living with human immunodeficiency virus (HIV) in the Dominican Republic and in other countries.

DETAILED DESCRIPTION:
OUTLINE:

Participants participate in three annual interviews and clinical exams that last approximately 2 hours. Study participants provide blood, urine, and swab samples from the cervix, anus, and vagina and receive a pelvic exam. Any positive results are followed up in the study clinic.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 25 - 49 years old will be eligible to participate in the study
* Women living with HIV who have an intact cervix
* Intent to reside in the Santo Domingo area
* Ability to attend routine study visits at IDCP for at least 24 months during the study. If women report that they anticipate relocating in the subsequent 24 months or anticipate difficulty attending study visits they will not be eligible
* Ability to understand the study timeline and procedures and the willingness to complete the informed consent process are also inclusion criteria

Exclusion Criteria:

* Women with a prior diagnosis of cervical cancer or a history of treatment for cervical precancerous lesions (CIN2+) will be excluded
* Women with significant physical, mental, or social conditions that would limit participation with study procedures will not be eligible for the study
* Women who are pregnant or report an intent to become pregnant in the subsequent 3 months will not be eligible for the study
* Women who have no history of vaginal sexual exposure will not be eligible for the study

Ages: 25 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 619 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Detection of cervical precancerous lesions (CIN2+) by cytology vs HPV restricted genotyping | At baseline
  Compare performance characteristics of two screening strategies. Comparison between dichotomous tests will be summarized by: (i) the true positive rate (TPR) and (ii) the false positive rate (FPR).

OTHER OUTCOMES:
Detection of CIN2+ is improved by cervical imaging with automated visual evaluation that uses a machine learning algorithm vs colposcopy | At baseline
  Post hoc evaluation not impacting treatment decision comparing colposcopy to image score by Cohen's kappa using a scale of normal, precancer+ and greyzone/low grade using a coordinated scale
Assess overall burden of HPV disease | At baseline
  Prevalence of non-cervical visible lesions, histological confirmation of non-cervix lesions (at the vulva, vagina, and peri-anal region), and hrHPV testing status at the vagina and anal canal
Detection of cervical precancerous lesions (CIN3) by cytology vs HPV restricted genotyping | At baseline
  Compare performance characteristics of two screening strategies. Comparison between dichotomous tests will be summarized by: (i) the true positive rate (TPR) and (ii) the false positive rate (FPR).
Cross-sectional diagnostic accuracy of triage by dual staining among hrHPV positive WLWH to detect CIN2+ | At baseline
  Estimate the diagnostic accuracy parameters (TPR, FPR, positive predictive value or PPV, negative predictive value or NPV) and their approximate 95% confidence intervals for the p16/Ki-67 dual staining triage strategy for WLWH who tested positive for restricted hrHPV genotyping at Month 0. Will also assess and compare the accuracy parameters (TPR/FPR) of the dual staining method as it applies to hrHPV16 positive WLWH versus those who are positive for other types of hrHPV in two-sample (unpaired) comparisons of proportions (two-sample proportion tests).
Diagnostic accuracy of dual staining triage among hrHPV positive WLWH to detect CIN2+ by specimen collected and reading approach | At baseline
  Calculate (i) the Cohen's kappa and (ii) the concordance correlation coefficient to calculate agreement between the two methods. Use the McNemar test to compare the overall agreement between them.
Diagnostic accuracy of hrHPV genotyping to detect CIN2+ among WLWH by vaginal vs cervical sampling | At baseline
  Calculate (i) the Cohen's kappa and (ii) the concordance correlation coefficient to calculate agreement between the two methods. Use the McNemar test to compare the overall agreement between them.
CIN2+ Incidence | At 12 and 24 months
  Estimate the cumulative incidence of newly detected CIN2+ over 2 years among women negative at previous time points.
Detection of repeat CIN2+ | At 12 and 24 months
  Calculate the proportion positive a second time for CIN2+ at Month 12 or 24.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret M. Madeleine, PhD, MPH, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Instituto Dermatológico Dominicano y Cirugía de Piel (IDCP) "Dr. Huberto Bogaert Diaz", Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: Yes
After publication of original data, data and specimens may be shared upon request with other investigators at academic or nonprofit institutions in a limited data set, as defined under HIPAA. The final dataset and specimens will be stripped of identifiers prior to release for sharing.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: One month after publication of the final report in manuscript form to a peer-reviewed journal.
Access Criteria: Investigators requesting access to data and specimens must sign a data-sharing agreement that provides for: (1) a commitment to using the data or specimens only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) not sharing the data or specimens with third parties. We reserve the right to limit data provided to outside investigators. We will not share data if we believe there is a possibility of deductive disclosure of subjects with unusual characteristics.

DOCUMENTS (1):
  • Informed Consent Form (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/72/NCT05556772/ICF_000.pdf